CLINICAL TRIAL: NCT06929910
Title: Evaluation of Systemic Therapy and the Effectiveness of Circulating Tumor DNA (ctDNA) Assays in Monitoring Treatment Response in Patients With Metastatic Cancer Undergoing K4Care Testing
Brief Title: Assessing Systemic Treatment and ctDNA Monitoring Efficacy in Metastatic Cancer Patients Using K4Care Testing.
Acronym: GS_ZKM
Status: Recruiting | Type: Observational
Sponsor: Gene Solutions (Industry)
Collaborators: The Medical Genetics Institute (MGI) of HCMC (Unknown)
Responsible Party: Sponsor
Other Study IDs: GS_ZKM
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Cancers
Keywords: ctDNA; metastatic cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to investigate the real-world treatment landscape of patients with metastatic cancer and determine the role of ctDNA in monitoring treatment response in patients with metastatic cancer who have undergone K4Care testing

DETAILED DESCRIPTION:
Study design: This is a prospective, longitudinal, non-interventional study. Samples will be collected from patients with metastatic cancer who have undergone K4Care testing at Gene Solutions from 03/2025 to 03/2026.

- Definition:

* Progression-free survival (PFS): The time from the start of treatment until disease progression, defined as the appearance of new tumor lesions or the spread of existing lesions to other organs or body parts.
* Overall survival (OS): The time from the start of the study (for non-randomized clinical trials) until death from any cause.
* Cell-free DNA (cfDNA) refers to DNA fragments released from cells into the bloodstream, with an average size of approximately 170 bp. A recent study showed that the concentration of cfDNA in the serum of cancer patients is elevated compared to healthy individuals. Circulating tumor DNA (ctDNA) refers to cfDNA released from cancer cells and carries tumor-associated mutations. The proportion of ctDNA within total cfDNA in cancer patients is highly variable, ranging from over 25% to as low as 0.01% (meaning that for every 10,000 cfDNA molecules in the blood, only 1 ctDNA molecule is released from cancer cells). This ratio is also known as the mutation allele fraction (MAF). MAF varies depending on the type and stage of cancer. The later the stage of the disease, the larger the tumor, and the more ctDNA is released into the blood. The presence of ctDNA in the serum indicates the presence of cancer in the body at the cellular level.

Due to the specificity of ctDNA for cancer, the correlation between ctDNA concentration and tumor size is less affected by other factors. Numerous studies have demonstrated that ctDNA levels change during treatment and correlate with early tumor response, which can be used as a companion biomarker and complement imaging response monitoring in patients treated with immunotherapy. Therefore, many studies have used ctDNA as a potential marker in monitoring tumor response in radical surgery, neoadjuvant chemoradiation, and evaluating treatment response in metastatic patients. NGS technology has brought tremendous value to the identification and treatment of cancer in recent years, helping to prolong the survival of patients and support the development of appropriate treatments for each patient with specific mutations. In addition, gene sequencing technology allows for the accurate detection of cancer-causing mutations in cfDNA samples, thereby identifying the composition of extracellular ctDNA released from the tumor.

* Blood sample: Each participant will have two times of 10mL blood sample collections, 1st blood sample collection is on the enrollment date and the 2nd blood sample collection is on the follow up visit date, from 3-6 months after the enrollment date or according to any participant follow-up visit during the study conduct.
* Clinical information to be collected: will be collected and supplemented (if missing) during the patient's follow-up visits as scheduled by the physician. The information to be collected includes:

  1. Basic patient demographics and medical history: age; sex; medical history (personal/family, viral infection status); diagnosis: time of diagnosis, cancer type (primary, secondary, metastatic), stage, location, histology, and other biochemical tests.
  2. Pathological results, immunohistochemical results, and biopsy site.
  3. Treatment regimen information: treatment types (surgery/chemotherapy/radiotherapy/targeted therapy), time points (start, mid-treatment, end of treatment):

     * Curative surgery
     * TKI/ICI or Chemotherapy for metastatic stage
     * Palliative treatment for metastatic stage
  4. Patient status: RECIST 1.1 response assessment at time points of Progressive Disease, Stable Disease, Partial Response, and Complete Response, based on the clinical physician's assessment documented in the medical record and accompanied by imaging (if available).

     * Time of progression and metastatic site
     * Survival status (alive or deceased). Cause of death. Time of death.
     * Information regarding death: the cause of death to evaluate whether it is related to cancer complications.
  5. Time of CT/MRI imaging, results, and clinical physician's interpretation (images can be provided if available)

ELIGIBILITY:
Inclusion Criteria:

* Pathological and imaging confirmation of metastatic or progressive stage IV cancer.
* Consent to the use of their clinical data.
* Diagnosis of one of the following common solid tumor types: lung, colorectal, breast, gastric, or cancer of unknown primary origin.
* Prior K4Care testing to identify tumor tissue (FFPE) mutations and consent to the use of their sequencing data.

Exclusion Criteria:

* Refusal to participate in the study.
* Absence of prior K4Care testing.
* Diagnosis of early-stage cancer or hematologic malignancy.
* Refusal to provide clinical information or blood samples.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic cancer who have had tumor tissue sequencing and have genetic mutation data from the K4Care test at Gene Solutions between [month/year] and [month/year], who consent to participate in the study and allow the use of their clinical and sequencing data for future research purposes, will be included. These patients will also receive free ctDNA monitoring using the K-Track N assay for 12 months.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
This study aims to evaluate the correlation between ctDNA clearance and treatment response in metastatic cancer: | 18 months
  * ctDNA clearance during and after treatment will reflect the patient's response to the treatment regimen.
  * Persistent positive ctDNA during and after treatment will reflect the patient's non-response to the treatment regimen and disease progression.
  According to current scientific reports, this correlation is independent of cancer type and treatment regimen. Moreover, this is a preliminary, observational, and descriptive statistical study. The sample size for each cancer type depends on the actual number of patients tested at Gene Solutions. Therefore, this study is not limited to a specific cancer type; all patients with metastatic cancer will be included in the analysis (similar to others design. With an average treatment response rate in the metastatic stage of 10-50%, a sample size of 200 patients will allow us to collect data for at least 20 patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Genetics Institute, Ho Chi Minh City, Hồ Chí Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data of this this study may be requested for publication by the journals, sharing anonymized data with suitable study will be decided by the sponsor, PIs and the authority agency where the data was collected. No identifiable information will be shared with any other person/organization than authority in the study.
Supporting Information: Study Protocol, ICF
Time Frame: Dec 2026
Access Criteria: GS_ZKM

REFERENCES:
- [Background] Kansara M, Bhardwaj N, Thavaneswaran S, Xu C, Lee JK, Chang LB, Madison RW, Lin F, Hsu E, Patel VK, Aleshin A, Oxnard GR, Simes J, Nimeiri H, Thomas DM. Early circulating tumor DNA dynamics as a pan-tumor biomarker for long-term clinical outcome in patients treated with durvalumab and tremelimumab. Mol Oncol. 2023 Feb;17(2):298-311. doi: 10.1002/1878-0261.13349. Epub 2022 Dec 13. PMID 36426653
- [Background] Bratman SV, Yang SYC, Iafolla MAJ, Liu Z, Hansen AR, Bedard PL, Lheureux S, Spreafico A, Razak AA, Shchegrova S, Louie M, Billings P, Zimmermann B, Sethi H, Aleshin A, Torti D, Marsh K, Eagles J, Cirlan I, Hanna Y, Clouthier DL, Lien SC, Ohashi PS, Xu W, Siu LL, Pugh TJ. Personalized circulating tumor DNA analysis as a predictive biomarker in solid tumor patients treated with pembrolizumab. Nat Cancer. 2020 Sep;1(9):873-881. doi: 10.1038/s43018-020-0096-5. Epub 2020 Aug 3. PMID 35121950
- [Background] Cabel L, Riva F, Servois V, Livartowski A, Daniel C, Rampanou A, Lantz O, Romano E, Milder M, Buecher B, Piperno-Neumann S, Bernard V, Baulande S, Bieche I, Pierga JY, Proudhon C, Bidard FC. Circulating tumor DNA changes for early monitoring of anti-PD1 immunotherapy: a proof-of-concept study. Ann Oncol. 2017 Aug 1;28(8):1996-2001. doi: 10.1093/annonc/mdx212. PMID 28459943
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Shuel SL. Targeted cancer therapies: Clinical pearls for primary care. Can Fam Physician. 2022 Jul;68(7):515-518. doi: 10.46747/cfp.6807515. No abstract available. PMID 35831091
- [Background] Kavun A, Veselovsky E, Lebedeva A, Belova E, Kuznetsova O, Yakushina V, Grigoreva T, Mileyko V, Fedyanin M, Ivanov M. Microsatellite Instability: A Review of Molecular Epidemiology and Implications for Immune Checkpoint Inhibitor Therapy. Cancers (Basel). 2023 Apr 13;15(8):2288. doi: 10.3390/cancers15082288. PMID 37190216
- [Background] Devarakonda S, Rotolo F, Tsao MS, Lanc I, Brambilla E, Masood A, Olaussen KA, Fulton R, Sakashita S, McLeer-Florin A, Ding K, Le Teuff G, Shepherd FA, Pignon JP, Graziano SL, Kratzke R, Soria JC, Seymour L, Govindan R, Michiels S. Tumor Mutation Burden as a Biomarker in Resected Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Oct 20;36(30):2995-3006. doi: 10.1200/JCO.2018.78.1963. Epub 2018 Aug 14. PMID 30106638
- [Background] Catalano M, Iannone LF, Nesi G, Nobili S, Mini E, Roviello G. Immunotherapy-related biomarkers: Confirmations and uncertainties. Crit Rev Oncol Hematol. 2023 Dec;192:104135. doi: 10.1016/j.critrevonc.2023.104135. Epub 2023 Sep 17. PMID 37717881
- [Background] Das S, Dey MK, Devireddy R, Gartia MR. Biomarkers in Cancer Detection, Diagnosis, and Prognosis. Sensors (Basel). 2023 Dec 20;24(1):37. doi: 10.3390/s24010037. PMID 38202898
- [Background] de Biase D, Fassan M, Malapelle U. Next-Generation Sequencing in Tumor Diagnosis and Treatment. Diagnostics (Basel). 2020 Nov 17;10(11):962. doi: 10.3390/diagnostics10110962. PMID 33212911
- [Background] Debela DT, Muzazu SG, Heraro KD, Ndalama MT, Mesele BW, Haile DC, Kitui SK, Manyazewal T. New approaches and procedures for cancer treatment: Current perspectives. SAGE Open Med. 2021 Aug 12;9:20503121211034366. doi: 10.1177/20503121211034366. eCollection 2021. PMID 34408877
- [Background] Anand U, Dey A, Chandel AKS, Sanyal R, Mishra A, Pandey DK, De Falco V, Upadhyay A, Kandimalla R, Chaudhary A, Dhanjal JK, Dewanjee S, Vallamkondu J, Perez de la Lastra JM. Cancer chemotherapy and beyond: Current status, drug candidates, associated risks and progress in targeted therapeutics. Genes Dis. 2022 Mar 18;10(4):1367-1401. doi: 10.1016/j.gendis.2022.02.007. eCollection 2023 Jul. PMID 37397557